CLINICAL TRIAL: NCT00487773
Title: Effect of Different Doses of Budesonide on Markers of Bone Metabolism in Children With Asthma - Randomized, Controlled Trial.
Brief Title: Effect of Different Doses of Budesonide on Markers of Bone Metabolism in Children With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Iwona Stelmach MD, PhD, Prof, Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: RNN-87-06-KE
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Asthma
Keywords: asthma; children; inhaled glucocorticosteroids; bone metabolism
MeSH Terms: conditions — Asthma | interventions — Budesonide; Cholecalciferol; montelukast; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): budesonide
  Interventions: Drug: budesonide
- 2 (Active Comparator): D3 vitamin
  Interventions: Drug: D3 vitamin
- 3 (Active Comparator): montelukast sodium
  Interventions: Drug: montelukast sodium
- 4 (Active Comparator): salbutamol
  Interventions: Drug: salbutamol

INTERVENTIONS:
Drug: budesonide — budesonide
  Arms: 1
Drug: D3 vitamin — D3 vitamin
  Arms: 2
Drug: montelukast sodium — montelukast sodium
  Arms: 3
Drug: salbutamol — salbutamol
  Arms: 4

SUMMARY:
The purpose of the trial is to check if inhaled glucocorticosteroids (iGCS) have influence on bone condition (if iGCS increases risk of osteoporosis and bone fraction) in children with asthma.

DETAILED DESCRIPTION:
Asthma is the most prevalent chronic disease of respiratory tract, the largest frequency is noticed in children. iGCS are the basic group of drugs in asthma, because of inflammatory character of disease. All iGCS are absorbed to the systemic circulation (small amounts) despite of local exposition in lungs and possess systemic effects. The purpose of trial is to check if iGCS have influence on bone condition (if iGCS increases risk of osteoporosis and bone fraction) in children with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Allergic only to house dust mites
* Never treated chronically (longer than at least 3 months) with anti-asthmatic drugs
* Newly-diagnosed or non-treated asthma
* Must be able to inhale drugs

Exclusion Criteria:

* Other allergic diseases requiring treatment with glucocorticosteroids
* Other chronic diseases
* Asthma exacerbation
* Pregnancy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Markers of bone metabolism (from serum and urine) | Baseline and 6 months

SECONDARY OUTCOMES:
Symptoms score (based on PAQLQ), spirometry | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Olszowiec-Chlebna, MD, Principal Investigator — Department of Pediatrics and Allergy, Medical University of Lodz, Poland; Iwona Stelmach, MD, PhD, Prof, Study Chair — Department of Pediatrics and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pediatrics and Allergy, Medical University of Lodz, Lodz, Poland